CLINICAL TRIAL: NCT01134367
Title: An Epidemiological, Postmarketing Observational Study to Describe Symptom Control and Impact of Gastroesophageal Reflux Disease (GERD) on Patients' Daily Life
Brief Title: An Epidemiological Study to Describe Symptom Control and Impact of Gastroesophageal Reflux Disease
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-GRS-DUM-2010/1
Record Dates: First submitted 2010-05-28; First posted 2010-06-02 (Estimated); Last update posted 2011-07-14 (Estimated); Status verified 2011-07

CONDITIONS: GERD
Keywords: gastroesophageal reflux disease (GERD)
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Patients with GERD

SUMMARY:
The purpose of this study is to examine patient's perspective of symptom control and impact of gastroesophageal reflux disease (GERD) on daily life.

ELIGIBILITY:
Inclusion Criteria:

* Patients with gastroesophageal reflux disease -GERD (disease duration ≤3 years or newly diagnosed) that are currently not treated with a proton pump inhibitor, for whom the general practitioner (GP) has previously decided to initiate or change the tre
* Patients should be treated for GERD according to current practice (National guideline for treatment of dyspepsia in GP setting)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinics
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Epidemiological data in a population of GERD patients with disease duration ≤ 3 years or newly diagnosed to include: Typical GERD symptoms (indicating frequency and severity of symptoms) and signs | 8 weeks
Epidemiological data in a population of GERD patients with disease duration ≤ 3 years or newly diagnosed to include: Demographic data | 8 weeks
Epidemiological data in a population of GERD patients with disease duration ≤ 3 years or newly diagnosed to include: Treatments for GERD and treatment changes | 8 weeks
Epidemiological data in a population of GERD patients with disease duration ≤ 3 years or newly diagnosed to include: Patient's perspective of symptom control and impact on daily life assessed using a patient-questionnaire (GIS-GERD Impact Scale). | 8 weeks

SECONDARY OUTCOMES:
To evaluate the added value of a patient questionnaire (GIS-GERD Impact Scale) as a useful tool for the initial and long-term management of GERD patients: determination of the appropriate treatment and evaluation of the response to treatment | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Miodrag Krstić, Prof.Dr, Principal Investigator — Institute for Gastroenterology, Clinical Center of Serbia, Belgrade; Dragomir Damjanov, Prof. Dr, Principal Investigator — Clinic for Internal Diseases, Clinical Center of Vojvodina, Novi Sad; Aleksandar Nagorni, Prof. Dr, Principal Investigator — Clinic for Internal Diseases- Gastroenterology Dept, Clinical Center Nis
Locations (7):
- Serbia (7):
  - Research Site, Belgrade
  - Research Site, Leskovac
  - Research Site, Niš
  - Research Site, Novi Sad
  - Research Site, Pančevo
  - Research Site, Subotica
  - Research Site, Zrenjanin